CLINICAL TRIAL: NCT03079830
Title: Efficacy of Ropivacaine Wound Infiltration for Postoperative Pain Management After Minimally Invasive Aortic Valve Surgery
Brief Title: Postoperative Pain Management After Minimally Invasive Aortic Valve Surgery
Acronym: PPMAMIAVS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Maja Sostaric, asoc. prof., University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KVIT2016
Record Dates: First submitted 2016-10-11; First posted 2017-03-15 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Aortic Valve Surgery; Postoperative; Pain
Keywords: aortic valve surgery; postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Pirinitramide; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ropivacaine continous infusion (Active Comparator): Piritramid
  Interventions: Drug: Piritramid
- Saline continous (Sham Comparator): Piritramid
  Interventions: Drug: Piritramid; Drug: Saline

INTERVENTIONS:
Drug: Piritramid — Piritramid will be administered i.v., if the patients feel pain after receiving a bolus of Ropivacaine or saline through the catheter.
  Other Names: Dipidolor
Drug: Saline — Piritramid will be administered i.v., if the patients feel pain after receiving a bolus of Ropivacaine or saline through the catheter.
  Other Names: Saline Solution
  Arms: Saline continous

SUMMARY:
The study evaluates the efficacy of local anesthestic application through the catheter in the surgical wound for the postoperative pain relief after minimally invasive aortic valve surgery. The patients will be enrolled in two different groups according to the protocol of the local anesthetic and saline administration:

1. group: continous infusion of the local anesthetic plus bolus on demand
2. group: continous infusion of saline plus bolus on demand For all patients metamizol every 12 hours plus bolous of piritramid on demand.

DETAILED DESCRIPTION:
Patients undergoing minimally invasive aortic valve replacment surgery will be enroled in the study, after giving a signed informed consent.

The study evaluates the efficacy of local anesthestic application through the catheter in the surgical wound for the postoperative pain relief after minimally invasive aortic valve surgery.

Patients will then be randomised in two groups according to the protocol:

1. group: continous infusion of the local anesthetic plus bolus on demand
2. group: continous infusion of saline plus bolus on demand

All patients will receive Metamizol every 12 hours plus bolus of piritramid on demand.

Analgesia effectivness will be checked hourly according to the visual analogue scale (VAS). According to protocol, bolus will be given every time the score of VAS scale is >3.

The catheter will be removed 48 hours after the protocols' start.

ELIGIBILITY:
Inclusion Criteria:

* Patients after minimally invasive aortic valve surgery
* Patients agreement with the study

Exclusion Criteria:

* Age under 18 years
* Allergy to local anesthetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-10; Primary Completion 2017-12-31 (Actual); Study Completion 2018-01-11 (Actual)

PRIMARY OUTCOMES:
Comparison of cumulative postoperative dose of Piritramid between the two different protocols, using VAS scale to determine level of analgesia. | 48 hours after admission to the intensive care unit (ICU)
  Comparison of cumulative postoperative dose of Piritramid between the two protocols

SECONDARY OUTCOMES:
Complications related to the catheter in the surgical wound | Up to 30 days
  Complications related to the catheter in the surgical wound
Visual analogue scale (VAS), frequency of scores higher than 3 | 48 hours after admission to the ICU
  Visual analogue scale (VAS), frequency of scores higher than 3
Patients satisfaction with pain relief measured by Likert-type Patient satisfaction scale | 72 hours after surgery
  Patients satisfaction regarding pain relief, in the following order 1.very satisfied 2.satisfied 3.neither satisfied nor dissatisfied 4.dissatisfied 5.completely dissatisfied
Rate of complications related to the local anesthetic | 72 hours after surgery
  Neurotoxicity and cardiotoxicity related to the local anesthetic
Hospital lenght of stay | Up to 30 days
  Hospital lenght of stay

CONTACTS AND LOCATIONS:
Overall Officials: Maja Sostaric, PhD, Study Chair — Clinical department of anesthesiology and intensive care
Locations (1):
- University Clinical Center Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mijovski G, Podbregar M, Ksela J, Jenko M, Sostaric M. Effectiveness of wound infusion of 0.2% ropivacaine by patient control analgesia pump after minithoracotomy aortic valve replacement: a randomized, double-blind, placebo-controlled trial. BMC Anesthesiol. 2020 Jul 18;20(1):172. doi: 10.1186/s12871-020-01093-9. PMID 32682395